CLINICAL TRIAL: NCT00322530
Title: Comparison of Dialysis Strategies in Critically Ill Patients With Acute Renal Failure on the Intensive Care Unit
Brief Title: Comparison of Dialysis Strategies in Critically Ill Patients With Acute Renal Failure
Acronym: rescue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Vedat Schwenger M.D, Prof. Dr. med., Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HD-Dialysis-2006
Record Dates: First submitted 2006-05-04; First posted 2006-05-08 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Dialysis; Acute Renal Failure
MeSH Terms: conditions — Acute Kidney Injury | interventions — Renal Replacement Therapy; Hybrid Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SLED (Active Comparator)
  Interventions: Procedure: Renal replacement therapy
- CVVHD (Active Comparator)
  Interventions: Procedure: Renal replacement therapy

INTERVENTIONS:
Procedure: Renal replacement therapy — ICU patients with acute renal failure were prospectively randomized to either CVVHD or SLED
  Other Names: sustained low efficiency dialysis (SLED); continous veno-venous hemodiafiltration (CVVHD)

SUMMARY:
The goal of the present study is the comparison of different dialysis strategies in critically ill patients with acute renal failure on the intensive care unit. Patients are treated with either continuous dialysis or hemofiltration. Outcome measures are death, restitution of renal function, days on ICU, hemodynamic stability, dialysis efficiency.

DETAILED DESCRIPTION:
The goal of the present study is the comparison of different renal replacement strategies in critically ill patients with acute renal failure on the intensive care unit. In a prospectively randomized clinical study patients are treated with either continuous dialysis (SLED) or continuous hemofiltration (CVVHD). 200 patients should be included in the study (n=100 each). The primary outcome is death at ICU, secondary outcome measures are restitution of renal function, days on ICU, hemodynamic stability, dialysis efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Written informed consent
* No pre-existing dialysis dependency

Exclusion Criteria:

* Minors / children
* No consent
* Severe electrolyte disturbances which necessitates special dialysis therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2006-04; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Death | 90 days

SECONDARY OUTCOMES:
costs | in hospital
Restitution of renal function | 90 days
days on ICU | in hospital
hemodynamic stability | in hospital
dialysis efficiency | in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Vedat Schwenger, MD, Principal Investigator — Division of Nephrology, University of Heidelberg
Locations (1):
- Division of Nephrology, University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Fayad AI, Buamscha DG, Ciapponi A. Timing of kidney replacement therapy initiation for acute kidney injury. Cochrane Database Syst Rev. 2022 Nov 23;11(11):CD010612. doi: 10.1002/14651858.CD010612.pub3. PMID 36416787
- [Derived] Tsujimoto Y, Miki S, Shimada H, Tsujimoto H, Yasuda H, Kataoka Y, Fujii T. Non-pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2021 Sep 14;9(9):CD013330. doi: 10.1002/14651858.CD013330.pub2. PMID 34519356
- [Derived] Schwenger V, Weigand MA, Hoffmann O, Dikow R, Kihm LP, Seckinger J, Miftari N, Schaier M, Hofer S, Haar C, Nawroth PP, Zeier M, Martin E, Morath C. Sustained low efficiency dialysis using a single-pass batch system in acute kidney injury - a randomized interventional trial: the REnal Replacement Therapy Study in Intensive Care Unit PatiEnts. Crit Care. 2012 Jul 27;16(4):R140. doi: 10.1186/cc11445. PMID 22839577